CLINICAL TRIAL: NCT07265765
Title: Effectiveness of Pilates Exercise in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Muhamed Kamal Omar, principal investigator (Physical Therapist), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pilates effect in shoulder SIS
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Subacromial Impingement Syndrome; Pilates Exercise; Shoulder Bursitis
Keywords: pilates exercise; subacromial impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Congresses as Topic; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator)
  Interventions: Behavioral: Conventional
- pilates exercise group (Experimental)
  Interventions: Behavioral: Pilates exercise

INTERVENTIONS:
Behavioral: Conventional — patients received conventional physical therapy exercise program that include (rotator cuff strength exercise, scapular stability exercise and posterior capsule stretch exercise) for 18 sessions for 6 weeks
  Arms: conventional group
Behavioral: Pilates exercise — patients who received the Pilates exercise in form of (shoulder drop, chest opener, book opening, scarecrow, dart, quadruped exercise, spine twist exercise).
  Arms: pilates exercise group

SUMMARY:
Subacromial Impingement Syndrome(SIS) is considered as one of the most common causes of shoulder pain, can be the source of considerable pain, disability and leads to limitations in activities of daily living.

This study aimed to investigate the effectiveness of the Pilates versus conventional treatment on shoulder pain, function, ROM and muscle strength in patients with SIS.

DETAILED DESCRIPTION:
Shoulder pain is the third most common chronic pain among musculoskeletal disorders, following low back pain and knee pain; it is usually characterized as non-traumatic complaints that arise from arm, neck and shoulder regions.

Approximately 50% of those experiencing shoulder pain have symptoms that indicate subacromial impingement syndrome (SIS) diagnosis; the prognosis varies widely; from pain to limited range of motion affecting their daily life activities: with about 40% of individuals suffer from pain one year later after their initial consulting with their primary care clinician.

The SIS is a painful condition that characterized by narrowing of the subacromial space that causes inflammation and degeneration of rotator cuff structures, resulting in pain during arm elevating.

Previous research identified many causes for the impingement such as poor posture, overuse or repetitive trauma, age-related changes, fatigue of the scapular and glenohumeral muscles, biomechanical alterations, neuromuscular adaptations, rotator cuff and deltoid muscle imbalances.

It leads to pain, disability, limited range of motion (ROM), loss of muscle strength, poor quality of life and sleep disturbances. There are many treatment approaches adopted for SIS such as conservative, pharmaceutical and surgical approach in severe cases.

Regarding the conservative it is considered the main treatment of SIS it often includes therapeutic exercises such as scapular stabilization exercises, rotator cuff strengthening exercises, stretching exercises and Pilates exercise that are effective in restoring shoulder function.

Pilates exercise was developed by Joseph Pilates as a comprehensive exercise, emphasizes the connection between mind and body control, making it a valuable tool in rehabilitation for enhancing core muscle strength, endurance, flexibility, posture, ROM, overall health, and quality of life are prevalent for both healthy individuals and rehabilitation purposes for SIS.

Pilates has been shown to effectively reduce shoulder pain, improve ROM, enhance posture, and support functional recovery in individuals with chronic shoulder pain, as highlighted in studies emphasizing its role in core stability and movement control even though it has a favorable impacts, the evidence to demonstrate its effect is limited.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 35-65 years old
* Presence of shoulder pain for at least three months
* Painful arc of movement during flexion or abduction or both
* The patient will be diagnosed with SIS if the tests of the Neer, Empty Can, and Hawkins will be positive during the physical examination.

Exclusion Criteria:

1. History of any surgical procedure to the affected upper extremity (Heron et al., 2017 and).
2. History of trauma, fracture, instability and shoulder dislocation to the shoulder in less than 12 weeks previously (EDA et al., 2016).
3. History of presence of cervical symptoms (neck pain, numbness or tingling in the upper extremity) (Heron et al., 2017).
4. History of corticosteroid injection in the shoulder region in the last 6 months (Turgut et al., 2017).
5. None- cooperative participants or cognitive impairment (a communication problem) (EDA et al., 2016).
6. History of any systemic illness, reflex sympathetic dystrophy and related syndromes e.g. rheumatoid arthritis, ankylosing spondylitis, diagnosed by physician (Heron et al., 2017 and Turgut et al., 2017).
7. Passive limitation of range of movement, stiff shoulder and less than 90 active elevation (Heron et al., 2017 and EDA et al., 2016).
8. Evidence of complete rotator cuff tear (positive drop arm test) (Heron et al., 2017).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
shoulder function | measured at baseline then after 6 weeks
  measured by the Arabic version of the SPADI (Shoulder Pain and Disability Index) is a self-report questionnaire designed to assess shoulder pain and disability in outpatients. It consists of 13 items: a 5-item pain subscale and an 8 item disability subscale; it is widely used and available in multiple languages such as the Arabic version ;with higher values indicating greater severity.
Shoulder Pian | at baseline and after 6 weeks
  measured using Numerical Pain scale It is a self-reported scale where the patient rates their pain on a numerical range, usually from 0 to 10; where the zero indicate less pain and 10 worst pain

SECONDARY OUTCOMES:
shoulder ROM(abduction and internal rotation) | measured at baseline and after 6 weeks
  measured by Digital goniometer The digital goniometer (DG)is a precise and user-friendly tool for measuring joint ROM in rehabilitation, offering real-time feedback and improved accuracy over the universal goniometer. It is commonly used for shoulder impingement assessment, helping track progress and ensures safe mobility improvements
shoulder muscle strength(UT,MT,LT,SA,ER,IR) | measured at baseline and after 6 weeks
  measured by HHD(Hand Held Dynamometer)(Lafayette) The handheld dynamometer (HHD) (model 01165, Lafayette Instrument Company, Indiana, USA)Is a reliable and objective tool for assessing isometric muscle strength, outperforming manual muscle testing. Lightweight and portable, it has strong concurrent validity, making it practical for strength evaluation. It is the preferred method for measuring shoulder rotator strength in symptomatic patients in clinical setting

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Alsanawi HA, Alghadir A, Anwer S, Roach KE, Alawaji A. Cross-cultural adaptation and psychometric properties of an Arabic version of the Shoulder Pain and Disability Index. Int J Rehabil Res. 2015 Sep;38(3):270-5. doi: 10.1097/MRR.0000000000000118. PMID 25954858
- [Result] Nazari G, MacDermid JC, Bryant D, Athwal GS. The effectiveness of surgical vs conservative interventions on pain and function in patients with shoulder impingement syndrome. A systematic review and meta-analysis. PLoS One. 2019 May 29;14(5):e0216961. doi: 10.1371/journal.pone.0216961. eCollection 2019. PMID 31141546
- [Result] Melo ASC, Moreira JS, Afreixo V, Moreira-Goncalves D, Donato H, Cruz EB, Vilas-Boas JP, Sousa ASP. Effectiveness of specific scapular therapeutic exercises in patients with shoulder pain: a systematic review with meta-analysis. JSES Rev Rep Tech. 2024 Jan 19;4(2):161-174. doi: 10.1016/j.xrrt.2023.12.006. eCollection 2024 May. PMID 38706660
- [Result] Lee SM, Lee CH, O'Sullivan D, Jung JH, Park JJ. Clinical effectiveness of a Pilates treatment for forward head posture. J Phys Ther Sci. 2016 Jul;28(7):2009-13. doi: 10.1589/jpts.28.2009. Epub 2016 Jul 29. PMID 27512253
- [Result] Desmeules F, Roy JS, Lafrance S, Charron M, Dube MO, Dupuis F, Beneciuk JM, Grimes J, Kim HM, Lamontagne M, McCreesh K, Shanley E, Vukobrat T, Michener LA. Rotator Cuff Tendinopathy Diagnosis, Nonsurgical Medical Care, and Rehabilitation: A Clinical Practice Guideline. J Orthop Sports Phys Ther. 2025 Apr;55(4):235-274. doi: 10.2519/jospt.2025.13182. PMID 40165544
- [Result] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Result] Chamorro C, Arancibia M, Trigo B, Arias-Poblete L, Jerez-Mayorga D. Absolute Reliability and Concurrent Validity of Hand-Held Dynamometry in Shoulder Rotator Strength Assessment: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Sep 3;18(17):9293. doi: 10.3390/ijerph18179293. PMID 34501883
- [Result] Byrnes K, Wu PJ, Whillier S. Is Pilates an effective rehabilitation tool? A systematic review. J Bodyw Mov Ther. 2018 Jan;22(1):192-202. doi: 10.1016/j.jbmt.2017.04.008. Epub 2017 Apr 26. PMID 29332746
- [Result] Atilgan E, Aytar A, Caglar A, Tigli AA, Arin G, Yapali G, Kisacik P, Berberoglu U, Sener HO, Unal E. The effects of Clinical Pilates exercises on patients with shoulder pain: A randomised clinical trial. J Bodyw Mov Ther. 2017 Oct;21(4):847-851. doi: 10.1016/j.jbmt.2017.02.003. Epub 2017 Mar 4. PMID 29037638
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32007452/